CLINICAL TRIAL: NCT05977374
Title: Effects of Low Impact Elliptical Training on Knee Osteoarthritis Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Collaborators: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Waqar Ahmed Awan, Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01238
Record Dates: First submitted 2023-07-11; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Masking Description: one of my groups is experimental and the other one is controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elliptical training group. (Experimental): In this group, Ultrasound 1MHz, 1.5W/cm2 7 mins, knee isometrics, and open chain activities. static stretching of the lower limbs will be given 10 reps each and held for 10 secs. 5 mins of warm-up activity on elliptical training will be given prior to the treatment group. then 3 mins of training with a set pace of 120 strides/min will start, then after 7 weeks, the timings will be increased to 5 mins. The base check-up will be conducted during 7 weeks and at the end of 12 weeks.
  Interventions: Other: experimental and conventional group
- Conventional treatment group (Other): Static stretching of the lower limbs as mentioned above, Ultrasound 1MHz 1.5W/cm2 7min, knee isometrics, open chain activities, anterior-posterior Maitland knee mobilizations grade 1 and 2, and home care plan.
  Interventions: Other: experimental and conventional group

INTERVENTIONS:
Other: experimental and conventional group — Static stretchings of the lower limb, Ultrasound 1 MHz 1.5W/cm2 7 mins, knee isometrics, open chain activities, knee mobilizations grade 1 and 2, and home care plan.
  Other Names: Conventional group

SUMMARY:
This research study is determined to see the effects of low-impact elliptical training on knee osteoarthritis outcomes.

DETAILED DESCRIPTION:
This study is designed to reduce the load of knee osteoarthritis patients in society so that the individual lives a healthy life without getting caught in any form of disability. Knee osteoarthritis is a progressive and degenerative disease of a joint that includes focal cartilage loss, bony hypertrophy, synovial capsule thickening, and changes in structures of periarticular ligaments and peripheral muscles.

There are several techniques used to overcome the individual's pain, for instance, the mobilization of the joint, prolotherapy, and the use of different electrical modalities. meanwhile, an elliptical workout provides a positive result in reducing the progression of overall knee joint and cartilage defects. elliptical training is included in low-impact activities which are proven joint-friendly activities for the better improvement of the knee joint.

This activity works on a similar principle of cyclic compressive loading as occurs in the manual mobilization of the knee joint. This activity brings out the fluid from the synovial membrane on compression and upon decompression, the cartilage reabsorbs the oxygen and nutrients, which crosses the synovial barrier into the synovial fluid through a double diffusion system in the joint. The fluid then reaches the extra-cellular matrix that moves to the multiple layers of chondrocytes for the growth of the cartilage in OA.

ELIGIBILITY:
Inclusion Criteria:

* 40- to 65-year-old.
* Diagnosed cases of Grade 1 and 2 Knee OA.
* Healthy and overweight patients will be included. (18.5- 29.5)

Exclusion Criteria:

* Acute musculoskeletal injury.
* Low back pain and Sciatica.
* Hip and ankle pathology.
* Acute infection, fever.
* The patient taking supplements and medications.
* Any knee deformity.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Knee joint pain. | Baseline, 6th week and 12th week.
  Pain is measured through KOOS questionnaire, which is the part of the KOOS and it has 9 items to identify pain scoring. A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
Knee joint X-rays. | Baseline, 6th week and 12th week.
  From the X-rays we will measure the medial and lateral knee joint space width through Radiant software.
Knee joint stiffness and symptoms. | Baseline, 6th week and 12th week.
  This is the part of KOOS questinnaire, it involves 5 items of symptoms and 2 items of stiffnss to rule out knee joint symptoms and stiffness. A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
Activities of daily livings impact on knee joint | Baseline, 6th week and 12th week.
  This is also the part of KOOS questionnaire, it includes 17 items to find out the scoring. A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
Sports activity impact on knee joint | Baseline, 6th week and 12th week.
  We can find the sports scoring through KOOS questionnaire, it embroils 5 items. A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
Quality of life impact on knee joint | Baseline, 6th week and 12th week.
  This one is also the part of KOOS questionnaire. it contain 4 items for scoring. A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.

CONTACTS AND LOCATIONS:
Locations (1):
- Islamabad Physical Therapy & Rehabilitation Centre, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No